CLINICAL TRIAL: NCT02970799
Title: Randomized, Controlled, Crossover Study Comparing Tear Production by Nasal Neurostimulation Versus Active Control
Brief Title: Tear Production by Nasal Neurostimulation Compared to Active Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oculeve, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: OCUN-016B
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Dry Eye; Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Intranasal then Extranasal Application (Experimental): Intranasal Neurostimulator applied intranasally (active) followed by extranasal application on Day 1. Participants were randomized to determine the intranasal and extranasal sequence for Days 15 and 29.
  Interventions: Device: Intranasal Neurostimulator
- Extranasal then Intranasal Application (Experimental): Intranasal Neurostimulator applied extranasally (control) followed by intranasal application on Day 1. Participants were randomized to determine the intranasal and extranasal sequence at Days 15 and 29.
  Interventions: Device: Intranasal Neurostimulator

INTERVENTIONS:
Device: Intranasal Neurostimulator — The device delivers small electrical currents, activating nerves that stimulate the body's natural tear production system.

SUMMARY:
This crossover design study evaluates the effectiveness of the Oculeve Intranasal Neurostimulator comparing the effect of intranasal (active) versus extranasal (control) stimulation on tear production as measured by the Jones Schirmer test in participants with dry eye disease.

DETAILED DESCRIPTION:
In this randomized, controlled study, participants will receive two applications of approximately a three-minute duration, one intranasal (active) and one extranasal (control), in randomized sequence at Visit 2 (Day 1). At Visits 3 (Day 15) and 4 (Day 29), participants will undergo two applications of approximately an eight-minute duration, one intranasal (active) and one extranasal (control), in randomized sequence. The Schirmer test is a clinically relevant and accepted measure to assess tear production over a specified time interval, generally five minutes. Tear meniscus height (TMH) and, to a lesser extent, tear meniscus area (TMA) have been reported as measures of tear quantity and/or production and have been used to diagnose dry eye disease (DED). One reliable means of measuring TMH and TMA is via use of optical coherence tomography (OCT), an established medical imaging technique that uses light to capture micrometer-resolution images from within optical scattering media such as biological tissue. Due to the non-invasive nature of the technique, this study was designed to explore the utility of TMH and TMA captured by OCT as a means of evaluating stimulated tear production following use of the study device.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe dry eye disease
* Have not worn contact lenses for at least seven days prior to the Screening Visit and willing to forego the use of contact lenses for the duration of the study
* Literate, able to speak English or Spanish, and able to complete questionnaires independently

Exclusion Criteria:

* Previously used the Intranasal Neurostimulator at any time
* Used commercial lid hygiene product within 14 days of the Screening Visit or plan to use at any time during the study
* Chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the investigator, may lead to the risk of clinically significant increased bleeding
* Nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
* Severe nasal airway obstruction (e.g. severe septal deviation or inferior turbinate hypertrophy) or vascularized polyp as confirmed by nasal endoscopic examination at the Screening Visit
* Have an implanted metallic or other electronic device in the head, a cardiac demand pacemaker, or an implanted defibrillator
* Participation in any clinical trial with a new active substance or a new device within 30 days of the Screening Visit

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Groups:
- Extranasal Then Intranasal Application: Intranasal Neurostimulator applied extranasally (control) on Day 1. Participants were randomized to determine the intranasal and extranasal sequence for Days 15 and 29.
Period: Overall Study
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Then Extranasal Application | Extranasal Then Intranasal Application | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Acute Tear Production by Jones Schirmer Test
Time Frame: Day 1
Population: as for baseline characteristics
Groups:
- Intranasal Application: Intranasal Neurostimulator applied intranasally (active) on Day 1 and Day 15 or 29.
- Extranasal Application: Intranasal Neurostimulator applied extranasally (control) on Day 1 and Day 15 or 29.
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Tear Meniscus Height
Time Frame: Pre and Post Application on Days 15 and 29
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Tear Meniscus Area
Time Frame: Pre and Post Application Days 15 and 29
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Number of Secreting Meibomian Glands
Time Frame: Day 1
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Tear Film Lipid Layer Thickness by Tearscope
Time Frame: Pre and Post Application on Days 15 and 29
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Lower Lid Margin Temperature
Time Frame: Pre and Post Application on Days 15 and 29
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Tear Film Temperature
Time Frame: Pre and Post Application on Days 15 and 29
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Adverse Events
Time Frame: Up to 41 days
Population: as for baseline characteristics
Arm/Group | Intranasal Application | Extranasal Application
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.
Arm/Group | Intranasal Application | Extranasal Application
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
During transfer and acquisition of study record by sponsors, no study data has been located and all efforts to locate study data have been exhausted. Therefore, no study data is available to report at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect cooperation among all parties involved in the study. Authorship will be established before writing the manuscript. The study sponsor and Ora will have the final decision regarding the manuscript and publication.